



F-CE-GEva-2C V1 (25.04.2019)

## **PATIENT INFORMATION SHEET**

| PROJECT TITLE: REBECCA - REsearch on BrEast Cancer induced chronic conditions | |
|---|---|
| supported by Causal Analysis of multi-source data | |
| STUDY TITLE: REBECCA-OST, Cancer-related osteopathy induced treatment | |
| https://rebeccaproject.eu/ | |
| PRINCIPAL INVESTIGATOR | Dr. Cristina Hernando Melià |
| SERVICE | Medical oncology |
| CENTER | University Clinical Hospital of Valencia |

We are writing to inform you about a research study in which you are invited to participate. The study has been approved by the Research Ethics Committee of its center, in accordance with current legislation, Law 14/2007, of July 3, on Biomedical Research. Our intention is that you receive the correct and sufficient information so that you can decide whether or not to agree to participate in this study. Read this information sheet carefully and we will clarify any doubts that may arise. In addition, you can consult with the people you consider appropriate. Likewise, you can request any explanation you want about any aspect of the study and its implications throughout it by contacting the principal investigator of the project, Dr. Hernando, on the phone 96 197 35 17.

# 1. Voluntary participation

We invite you to participate in the study because you have been prescribed an aromatase inhibitor treatment, following the usual clinical practice in the treatment of your disease.

You should know that your participation in this study is voluntary and that you may CHOOSE NOT to participate. If you choose to participate, you can change your decision and withdraw consent at any time, without altering your relationship with your doctor or causing any harm to your health care.

# 2. Justification and Objective of the study

This study aims to explore the potential of "real-world data" as a tool for monitoring patients treated with aromatase inhibitor. Real-world data informs about people's behaviors and routines, and is collected through mobile devices and apps.

The objective of this study is to check if there is a relationship between bone density levels and certain functional and emotional indicators of patients (extracted from "real-world data"), so that the analysis of dich to information allows to detect people at high risk of fracture.

# 3. Description of the study

This study will be carried out at the University Clinical Hospital of Valencia, and it is expected that 82 patients aged between **18 and 75 years**, **diagnosed with breast cancer** (stages I, II or III), and who are going to start or have started in the last 12 months, treatment with **aromatase inhibitor**, within routine clinical practice.





F-CE-GEva-2C V1 (25.04.2019)

The patients will be divided into two groups (41 patients for each of them) according to their bone density:

- 1. Group "Normal densitometry mild osteopenia": if the result of densitometry is greater than -1.5.
- 2. Group "Severe osteopenia Osteoporosis": if the result is less than or equal to -1.5.

You should know that bone densitometry is a non-invasive, painful, X-ray-like test performed on patients receiving aromatase inhibitor treatment before starting their treatment, following standard clinical practice.

The study aims to **collect information from patients through** the use of **mobile devices and applications** (on lifestyle habits, Internet use, emotional state, quality of life and satisfaction with treatment), **thus complementing the data collected during medical visits established by** routine clinical practice. Clinical information is collected internally through the use of a clinical registration form, while supplementary information is collected through the use of:

- an activity bracelet, also called a smartwatch;
- a computer application designed for the patient (pApp);
- optionally, a computer application designed for the figure of the partner<sup>1</sup> (cApp).
- A complementary program of the patient's Internet browser.

## What information will each of these devices collect?

The **activity tracker** or smartwatch captures, through sensors, data from: acceleration, heart rate, heart rate variation, heart rate during sleep, blood oxygen saturation level, number of steps, stress (based on heart rate information and heart rate variation), time and quality of sleep, intensity of movement/physical activity... This activity bracelet connects exclusively and directly, via *Bluetooth* technology, with the patient computer application (pApp), installed on your mobile phone, to transfer the recorded data.

## The patient computing application (pApp):

- connects with the activity tracker and recovers the captured data;
- collects the location signal (GPS) of the mobile phone;
- samples and makes available to the patient brief questionnaires (approximately 2-8 questions) to collect information on fatigue, mood, lifestyle habits;
- It allows the patient, if desired, to take photographs from the application itself<sup>2</sup> and make annotations about them (thus providing information, for example, about their diet or their environment).

\_

<sup>&</sup>lt;sup>1</sup> The partner is a **person chosen by The patient** to provide information on his activity Environment and state, belonging to the closest environment of <u>The patient</u>.

<sup>&</sup>lt;sup>2</sup> Only the **Photographs that the patient wants to take from the application** (Papp) shall be used in the study. This excludes photos taken from outside the app (e.g. from your mobile phone's camera).





F-CE-GEva-2C V1 (25.04.2019)

The **partner's computer application (cApp)** has brief questionnaires on quality of life, symptoms or close environment of the patient, to which the colleague responds. The use of this application is optional, always in the event that the patient wishes to designate a person she trusts with whom she shares her environment.

The browser add-on program is installed on the patient's computer and collects data on Internet usage. At any time, the patient can stop and resume monitoring her activity. Likewise, you can delete any data that you do not want to provide. In any case, all data will be pseudonymised, <sup>3</sup>since no personally identifiable information is collected (name, IP ...) and patients are characterized by a unique code. The data captured by this browser add-on is:

- Web pages visited: address, page name, user, time of visit.
- Search terms entered in Internet search engines.
- Activity on platforms and social networks (Facebook, Youtube, Instagram ...) including: shortcuts, pages and titles of conversations, search terms, visits made (user, time of visit in profiles or groups of a certain social network or platform), comments, reactions to comments from third parties (me like, dislike, emoticons, etc.).

# 4. Study activities

The present study lasts approximately 12 months. At the start of the study all participants, regardless of group, as well as a person of their choice, will be trained in the use of the REBECCA system, which includes mobile devices and apps, and an online tracking platform. Each participant, as well as the person he has designated, will provide through this system information of interest about his daily life, which requires an approximate dedication of between 15 and 30 minutes a day to respond to application notices and questionnaires. The REBECCA system will allow the collection of information throughout the study on the patient's lifestyle habits, the use she makes of the Internet, as well as her mood and quality of life.

Following standard clinical practice in individuals receiving aromatase inhibitor therapy, patients will attend two follow-up check-ups, at 6 and 12 months, to assess treatment progress and adherence, and will undergo densitometry at 12 months.

As a result of participating in this study, patients will undergo <u>additional densitometry at</u> <u>6 months</u>. This additional test will be coincided as much as possible with routine appointments, to minimize travel.

## 5. Risks and inconvenience arising from your participation in the study

Your participation in the study involves regular use of mobile devices and apps that allow the collection of data on their lifestyle habits, Internet use, mood and quality of life. The mobile device that will be used during the study is an activity bracelet, such as those commonly used during sports. The use of these bracelets does not pose any risk. However, it

HIP/CI V.0 05/01/22

<sup>&</sup>lt;sup>3</sup> The datos ppseudonymised do not allow identify directly to the individuals from whom they come.





F-CE-GEva-2C V1 (25.04.2019)

should be borne in mind that the use of applications requires interaction time (attending notices, answering questionnaires) and that the use of the mobile device involves wearing the bracelet correctly placed around the wrist.

#### 6. Possible benefits

Itis quite possible that you will not obtain any benefit in the prognosis and treatment of breast cancer by participating in this study, however, it could help prevent osteopenia and osteoporosis induced by adjuvant treatment of breast cancer with aromatase inhibitor in future patients.

## 7. Protection of personal data

The researcher and the center are respectively responsible for the processing of their data and undertake to comply with the data protection regulations in force, Organic Law 3/2018, of December 5, on the Protection of Personal Data and Guarantee of Digital Rights and Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016 on Data Protection (RGPD).

The data collected for the study will be identified by a code, so that it does not include information that can identify you, and only your doctor/collaborators could relate this data to you and your medical history. Therefore, your identity will not be revealed to any person except for exceptions in case of medical emergency or legal requirement.

Access to your personally identified information will be restricted to the study physician/collaborators, competent authorities, the Research Ethics Committee and personnel authorized by the sponsor (study monitors, auditors), when they need it to verify the data and procedures of the study, but always maintaining the confidentiality of the same in accordance with current legislation.

In accordance with the provisions of data protection legislation, you can exercise the rights of access, modification, opposition and cancellation of data, for which you must contact your study doctor. If you decide to withdraw consent to participate in this study, no new data will be added to the database, but those that have already been collected will be used.

In addition, you can limit the processing of data that is incorrect, request a copy or that the data you have provided for the study is transferred to a third party (portability). To exercise your rights, contact the principal investigator of the study or the Data Protection Officer of the center/institution in dpd@gva.es. You also have the right to contact the Data Protection Agency if you are not satisfied.

The encrypted data may be transmitted to other countries of the European Union, but in no case will they contain information that can directly identify you, such as name and surname, initials, address, social security number, etc. In the event that this transfer occurs, it will be for the same purposes of the study described or for use in scientific publications, but always maintaining the confidentiality of the same in accordance with current legislation.





F-CE-GEva-2C V1 (25.04.2019)

The researcher will take the appropriate measures to ensure the protection of your privacy and will not allow your data to cross with other databases that could allow your identification. If the investigator cannot confirm this claim, the patient should be informed of the risk of reidentification arising from the reuse of their data in future studies not defined at this time.

# 8. INFORMATION CONCERNING BIOLOGICAL SAMPLES

Their participation in this study <u>does not involve the collection and use of biological samples for research purposes.</u>





F-CE-GEva-2C V1 (25.04.2019)

# **INFORMED CONSENT**

| | INI ONNED CONSENT |
|---|---|
| PROJECT TITLE: REBECCA - REsearch on BrEast Cancer induced chronic conditions | |
| supported by Causal Analysis of multi-source data | |
| STUDY TITLE: REBECCA-OST, | Cancer-related osteopathy induced treatment |
| STUDY CODE | |
| PRINCIPAL INVESTIGATOR | Dr. Cristina Hernando Melià. |
| SERVICE | Medical oncology. |
| CENTER | University Clinical Hospital of Valencia |
| I understand that my participation I understand that I can withdraw fr -Whenever Without having to give explanation - Without this affecting my medical I freely agree to participate in the | given to me about the study. about the study. on about the study. written name by the patient) is voluntary. rom the studio: ons. al care. study. ssing of my personal data for this investigation under the |
| I will receive a signed and dated of Participant's signature | copy of this informed consent document Researcher's signature |
| Date://<br>(signature and handwritten date b | Date://<br>y the patient) |





F-CE-GEva-2C V1 (25.04.2019)

# **INFORMED CONSENT LEGAL REPRESENTATIVE**

| PROJECT TITLE: REBECCA - F | REsearch on BrEast Cancer induced chronic conditions |
|---|---|
| supported by Causal Analysis | of multi-source data |
| STUDY TITLE: REBECCA-OST | , Cancer-related osteopathy induced treatment |
| STUDY CODE | |
| PRINCIPAL INVESTIGATOR | Dr. Cristina Hernando Melià. |
| SERVICE | Medical oncology. |
| CENTER | University Clinical Hospital of Valencia |
| I,>><<_ | |
| (Handwritten name by repres | sentative) |
| as>><< | |
| >><<_ | |
| (Handwritten name by repres | |
| I have read the information sheet | • |
| I have been able to ask questions | • |
| I have received enough information | on about the study. |
| I have spoken to>>< | and the angle of the control of the |
| • | name by representative) |
| I understand that your participatio | · |
| I understand that you can withdra | w from the study: |
| -Whenever. | |
| - Without having to give explanation | |
| - Without this affecting your medic | cal care. |
| I freely consent to your participation | • |
| • | sing of your personal data for this investigation under the |
| conditions explained in this inform | nation sheet. |
| • | ed copy of this informed consent document |
| Signature of the legal representation | • |
| member or de facto related perso | n |
| | _ , |
| Date:// | Date:/ |
| (Signature and handwritten | date by the |
| representative) | |





F-CE-GEva-2C V1 (25.04.2019)

# **INFORMED CONSENT TO WITNESSES**

| | RESearch on Breast Cancer Induced Chronic Conditions |
|---|---|
| supported by Causal Analysis | , Cancer-related osteopathy induced treatment |
| STUDY CODE | , Cancer-related Osteopathy induced treatment |
| PRINCIPAL INVESTIGATOR | Dr. Cristina Hernando Melià. |
| SERVICE | Medical oncology. |
| CENTER | University Clinical Hospital of Valencia |
| You have been able to ask questing You have received enough informing You have spoken with >><< (Hand You understand that your participation of you understand that you can with the work of th | o you about the study has been read, so that: ons about the study. nation about the study. dwritten name by witness) ation is voluntary. draw from the study: ons. cal care. ation in the study. essing of your personal data for this investigation under the |
| You will receive a signed and date Signature of the witness Date:// | ed copy of this informed consent document Researcher's signature Date:// |
| (Signature and handwritten date b | by the witness |